CLINICAL TRIAL: NCT01621204
Title: Treatment of thromBocytopenia With EltRombopag or Intravenous Immune Globulin (IVIG) Before and DurING Invasive Procedures in Patients With Immune ThrombocytoPenia- BRIDGING ITP Study
Brief Title: A Trial of Eltrombopag or Intravenous Immune Globulin Before Surgery for Immune Thrombocytopenia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: GlaxoSmithKline (Industry); Hamilton Health Sciences Corporation (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Donald Arnold, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M-EIBS-A-12
Record Dates: First submitted 2012-06-12; First posted 2012-06-18 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Thrombocytopenia; ITP; Platelets; Bleeding; Immune; Eltrombopag; IVIG
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Hemorrhage | interventions — eltrombopag; Immunoglobulins, Intravenous; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eltrombopag (Experimental): Eltrombopag is a small molecule, non-peptide thrombopoietin (TPO) receptor agonist indicated for the treatment of thrombocytopenia in patients with chronic ITP who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy. TPO receptor agonists are an effective new class of medications that are non-immunogenic agonists of the TPO receptor (c-Mpl) and work by increasing platelet production in ITP patients.
  Interventions: Drug: Eltrombopag
- IVIG infusion (Active Comparator): Intravenous immunoglobulin (IVIG) is used to rapidly increase platelet counts in ITP patients. IVIG is associated with a transient platelet count response in approximately 80% of patients, which occurs within 2 - 4 days. It is commonly used to improve platelet count numbers prior to surgery for patients with ITP.
  Interventions: Drug: IVIG infusion

INTERVENTIONS:
Drug: Eltrombopag — Participants are started on 50mg daily oral pill (or 25mg daily for patients of East Asian descent) 21 days before surgery. Dose may be adjusted based on subsequent platelet counts (minimum 25mg; maximum 75mg).
  Other Names: Revolade
  Arms: Eltrombopag
Drug: IVIG infusion — IVIG infusion (1-2 g/kg) given 7 (+/-2) days prior to surgery; with an additional infusion allowed within one week of achievement of surgical hemostasis, if needed
  Other Names: Intravenous Immunoglobulin; IgG
  Arms: IVIG infusion

SUMMARY:
This is a study to investigate if eltrombopag can be used instead of Intravenous Immune Globulin (IVIG) in patients with ITP, to adequately raise their platelet count when they undergo minor or major surgery. Eltrombopag is a daily, oral pill approved for treatment of ITP. IVIG is a blood product frequently used to treat ITP. Patients with ITP who need surgery have to get treatment to increase their platelet count. IVIG is commonly used for this purpose but eltrombopag may be more effective and convenient for patients.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a heterogeneous autoimmune disease characterized by the presence of platelet autoantibodies, low platelet counts and an increased risk of bleeding. TPO receptor agonists which stimulate platelet production have been shown to be remarkably effective in ITP. Their use as a short-term means of elevating platelet counts in preparation for surgical procedures has not yet been adequately evaluated.

Many patients with moderate to severe ITP (platelet count less than 50 x 10exp9/L) have stable platelet counts and do not bleed; however, when surgeries or invasive procedures become necessary, additional treatment is often required to increase the platelet count to achieve adequate hemostasis. Although specific guidelines for surgical platelet count thresholds in ITP are lacking, platelet transfusion guidelines recommend a platelet count of 50 - 100 x10exp9/L for the vast majority of surgical procedure; 50x10exp9/L is a typical threshold for minor surgeries like tooth extractions and endoscopies; and 100x10exp9/L is used for major surgery like cardiac surgery or neurosurgery.

Commonly, intravenous immunoglobulin (IVIG) is used to rapidly increase platelet counts in ITP patients before an invasive procedure. IVIG is associated with a transient platelet count response in approximately 80% of patients, which occurs within 2 - 4 days. In most patients, platelet counts remain elevated for approximately 4 weeks, allowing enough time to complete the procedure and for adequate post-operative hemostasis. However, IVIG is a resource-intensive and expensive blood product associated with frequent side effects.

Eltrombopag is a small molecule, non-peptide thrombopoietin (TPO) receptor agonist indicated for the treatment of thrombocytopenia in patients with chronic ITP who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy. TPO receptor agonists are an effective new class of medications that are non-immunogenic agonists of the TPO receptor (c-Mpl) and work by increasing platelet production in ITP patients. In randomized controlled trials, eltrombopag maintenance therapy has been shown to raise the platelet count in 60 - 80% of ITP patients and platelet counts generally remain elevated as long as the drug is continued. Time to response is 1 - 2 weeks with minimal need for dose titration. Side effects of eltrombopag observed in clinical studies included elevation of liver enzymes (approximately 10% of patients). The risk of thrombosis and bone marrow reticulin formation remain uncertain.

The investigators propose a randomized controlled trial (RCT) involving 74 patients (across approximately 8 centers) in Canada. This study will evaluate the efficacy and safety of eltrombopag bridging therapy compared with IVIG bridging therapy in adult patients with ITP who require surgery. This study will also evaluate bleeding, adverse events and patient-reported treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM). Patients will be stratified according to centre and surgery type (major vs. minor).

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary ITP;
* Platelet count below surgical platelet count threshold (50 x10^9/L for minor surgery; 100 x 10^9/L for major surgery);
* 18 years of age or older;
* On stable doses of concomitant ITP medications (i.e the dose administered has not changed) or no ITP medication for at least 2 weeks;
* At least 3-weeks lead time available between randomization and scheduled surgery;
* IVIG and Eltrombopag are acceptable ITP treatment options for this patient;
* Able to provide informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Treatment with IVIG within the last 2 weeks;
* Treatment with a thrombopoietin receptor agonist (eltrombopag or romiplostim) within the last 4 weeks;
* AST, ALT above 2X upper limit of normal;
* Bilirubin above 1.5X upper limit of normal in the absence of clinically benign liver disorder (eg. Gilberts syndrome);
* Deep vein thrombosis, myocardial infarction, thrombotic stroke or arterial thrombosis in the last 12 months;
* History of bone marrow reticulin or fibrosis;
* Known liver cirrhosis;
* Active malignancy (defined as requiring treatment or palliation within the last 6 months);
* Any additional laboratory test result, health related illness or other diagnosis which, in the opinion of the treating physician, may put the subject's health or safety at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Achievement of a platelet count level that is above the platelet count threshold for surgery preoperatively and that is maintained above the threshold during the post-hemostasis period without the use of rescue treatment | For a the period of time from the final pre-operative visit until 7 days after surgical hemostasis is achieved
  Threshold is a platelet count of 50 x 10^9/L for minor surgery and 100 x 10^9/L for major surgery.

SECONDARY OUTCOMES:
Time to treatment failure | During the period from the final pre-operative visit until 7 days after surgical hemostasis is achieved
  Time to the occurrence of a platelet count level below the designated threshold, or the administration of rescue treatment
Surgical delays or cancellations | Measured at time of planned surgery
  Proportion of patients with surgical delays or cancellations
Bleeding | During treatment and follow up (on average, 8 weeks from starting treatment)
  Graded as per the ITP bleeding score
Thrombocytosis | During treatment and follow up (on average, 8 weeks from starting treatment)
  Platelet count >400 x 10^9/L
Blood product transfusions | During treatment and follow up (on average, 8 weeks from starting treatment)
  Proportion of patients requiring platelet, red blood cells and plasma transfusions
Rescue treatment | During the period from the final pre-operative visit until 7 days after surgical hemostasis is achieved
  New ITP treatment (typically platelet transfusions, high dose IVIG or high dose corticosteroids) or an increased dose of existing ITP treatment administered to increase platelet counts above threshold
Platelet count change over time | During treatment and follow up (on average, 8 weeks from starting treatment)
  Trend of all platelet count measurements in the trial
Patient satisfaction with treatment | Immediately before surgery (final pre-op visit) and 7 days (+/- 2 days) after surgical hemostasis is achieved
  Assessed using the Treatment Satisfaction Questionnaire for Medications Score vII (which incorporates effectiveness, convenience, side effects, and overall satisfaction)
Hospitalizations | During treatment and follow up (on average, 8 weeks from starting treatment)
  Unanticipated admissions to hospital or prolongation of hospitalization
Thrombosis | During treatment and follow up (on average, 8 weeks from starting treatment)
  Symptomatic thrombotic events confirmed with diagnostic imaging
Adverse Events | During treatment and follow up (on average, 8 weeks from starting treatment)
  Defined using the Common Terminology Criteria for Adverse Events v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Arnold, MD MSc, Principal Investigator — McMaster University
Locations (10):
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - St.Micheal's Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- The Haga Hospital, The Hague, Netherlands

REFERENCES:
- [Result] Arnold DM, Heddle NM, Cook RJ, Hsia C, Blostein M, Jamula E, Sholzberg M, Lin Y, Kassis J, Larratt L, Tinmouth A, Amini S, Schipperus M, Lim W, Vishnu P, Warner M, Carruthers J, Li N, Lane S, Kelton JG. Perioperative oral eltrombopag versus intravenous immunoglobulin in patients with immune thrombocytopenia: a non-inferiority, multicentre, randomised trial. Lancet Haematol. 2020 Sep;7(9):e640-e648. doi: 10.1016/S2352-3026(20)30227-1. PMID 32853584
- [Derived] Arnold DM, Jamula E, Heddle NM, Cook RJ, Hsia C, Sholzberg M, Lin Y, Kassis J, Blostein M, Larratt L, Amini S, Schipperus M, Carruthers J, Lane SJ, Li N, Kelton JG. Peri-Operative Eltrombopag or Immune Globulin for Patients with Immune Thrombocytopaenia (The Bridging ITP Trial): Methods and Rationale. Thromb Haemost. 2019 Mar;119(3):500-507. doi: 10.1055/s-0038-1677531. Epub 2019 Jan 27. PMID 30685874